CLINICAL TRIAL: NCT03381794
Title: Trends in Corneal Transplantation from 2001 in Germany: Reports of the DOG-Section Cornea and Its Keratoplasty Registry
Brief Title: The German Keratoplasty Registry of the German Ophthalmological Society (DOG)
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Collaborators: University Eye Hospital, Freiburg (Other); University of Erlangen-Nürnberg (Other); University of Cologne (Other); Heinrich-Heine University, Duesseldorf (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Elias Flockerzi, Principal Investigator, Resident of Ophthalmology, University Hospital, Saarland
Other Study IDs: GeKeR
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Corneal Transplantation
Keywords: Keratoplasty Registry, PKP, DSAEK, DMEK, DALK
MeSH Terms: interventions — Corneal Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 16 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with corneal transplantation: Aim is to include all patients in Germany treated with the different types of corneal transplantation.
  Interventions: Procedure: Corneal transplantation

INTERVENTIONS:
Procedure: Corneal transplantation — PKP: Penetrating Keratoplasty DALK: Deep Anterior Lamellar Keratoplasty DMEK: Descemet Membrane Endothelial Keratoplasty DSAEK: Descemet's Stripping Automated Endothelial Keratoplasty
  Other Names: PKP, DALK, DMEK, DSAEK

SUMMARY:
Aim of this study is to reflect on the changing trends in absolute numbers, surgical techniques and indications of corneal transplantations being performed in Germany.

The Section Cornea of the German Ophthalmological Society provides interim-assessments on a regular basis about the most up-to-date results of this long-term study.

ELIGIBILITY:
Inclusion Criteria:

All patients in Germany treated with the different types of corneal transplantation since 2001.

Exclusion Criteria:

Patients without corneal transplantation.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Germany treated with the different types of corneal transplantation since 2001.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
An overview about absolute numbers of corneal transplantation in Germany. | 01/01/2001 to 31/12/2031
  A questionnaire about absolute numbers of corneal transplantation per year was sent to the 111 ophthalmological departments in Germany performing corneal transplantation. Data has been and is collected annually since 2001.
An overview about trends in the various types of corneal transplantation in Germany. | 01/01/2001 to 31/12/2031
  The questionnaire also records the types of corneal transplantation (i.e. penetrating keratoplasty, deep anterior lamellar keratoplasty, Descemet membrane endothelial keratoplasty (DMEK) and Descemet's stripping automated endothelial keratoplasty DSAEK) allowing a discussion of trends in corneal transplantation. Data has been and is collected annually since 2001.
An overview about indications for corneal transplantation in Germany. | 01/01/2001 to 31/12/2031
  The questionnaire also records the indications for corneal transplantation (e.g. Fuchs' endothelial corneal dystrophy, pseudophakic corneal decompensation, repeated keratoplasty after graft failure, keratoconus and corneal scarring). Data has been and is collected annually since 2001.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Seitz, Prof.Dr.med., Study Director — Universität des Saarlandes
Locations (1):
- Department of Ophthalmology, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flockerzi E, Turner C, Seitz B, Collaborators GSG; GeKeR Study Group. Descemet's membrane endothelial keratoplasty is the predominant keratoplasty procedure in Germany since 2016: a report of the DOG-section cornea and its keratoplasty registry. Br J Ophthalmol. 2024 May 21;108(5):646-653. doi: 10.1136/bjo-2022-323162. PMID 37586835
- [Background] Flockerzi E, Maier P, Bohringer D, Reinshagen H, Kruse F, Cursiefen C, Reinhard T, Geerling G, Torun N, Seitz B; all German Keratoplasty Registry Contributors. Trends in Corneal Transplantation from 2001 to 2016 in Germany: A Report of the DOG-Section Cornea and its Keratoplasty Registry. Am J Ophthalmol. 2018 Apr;188:91-98. doi: 10.1016/j.ajo.2018.01.018. Epub 2018 Feb 2. PMID 29410297